

## **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

| Integrating acupuncture into posundergoing open abdominal opera 2020-0234 | • | management | in | patients |
|---|---|---|---|---|
| Study Chair: Wenli Liu, M.D. | | | | |
| Participant's Name | Medical Record N | lumber | _ | |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

#### STUDY SUMMARY

The goal of this research study is to learn if it is possible to use acupuncture after surgery in patients who are having open colorectal or pancreatic surgery. Researchers want to learn if acupuncture may help to reduce after-surgery side effects and improve recovery.

This is an investigational study. Acupuncture needles are an FDA approved medical device, but acupuncture therapy itself is considered investigational. It is investigational to use acupuncture in an attempt to improve recovery after colorectal or pancreatic surgery.

Acupuncture may help to reduce post-operative symptoms including pain. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. If you take part in this study, you may experience discomfort or pain due to treatment, including aching at the acupuncture site, and/or pain or discomfort from the other study procedures. Questionnaires may include uncomfortable questions.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You will receive daily acupuncture treatment for up to 7 days if you are assigned to the acupuncture arm, starting on the day after your surgery. The study period starts the day after surgery and ends when you are discharged from the hospital.

The study will be performed at no cost to you. You and/or your insurance provider will still be responsible for the costs of surgery and hospitalization.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive other investigational therapy, if available. Pain management is part of the post-operative care for this study. In all cases, you will receive appropriate medical care, including treatment for pain.

## 1. STUDY DETAILS

Up to 70 patients will be enrolled in this study. All will take part at MD Anderson.

If you agree to take part in this study, information from your medical record (such as your age, weight/height, your medical history, cancer stage, the type of procedure that is performed and your post-operative recovery, the results of any laboratory tests, and symptoms you may be experiencing) will be collected and stored in a research database.

The acupuncture sessions are 1 time a day for up to 7 days. The acupuncture treatments are provided by 3 board-certified acupuncturists who have been credentialed by the MD Anderson Credentialing Office. Each acupuncture session will take about 25 minutes. In each acupuncture session, very small, sterile needles made of stainless steel will be inserted and removed from specific points on the body for the purpose of reducing your sensation of post-operative symptoms including pain. Acupuncture needles may be stimulated manually or electronically to improve treatment effects.

You will be asked to complete questionnaires about symptoms and pain at the time of consent, on the day after surgery, and then right after your acupuncture session every 2 days. These will take about 10 minutes each time.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

**Acupuncture** may cause a tingling sensation and/or an ache around the needles. It may cause redness, infection, fainting, and/or bruising at the acupuncture site. It may also cause an allergic reaction, including skin inflammation from the stainless steel and swelling of the arms and torso. If you feel uncomfortable at any time, you may ask to have the acupuncture stopped.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns after completing the questionnaire(s), you are encouraged to contact your doctor or the study chair. There are no plans to provide you compensation from such developments.

This research is covered by a Certificate of Confidentiality (CoC) from the National Institutes of Health. The researchers with this CoC may not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information protected by this CoC cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below).

The CoC cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation. You should understand that a CoC does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The CoC will not be used to prevent disclosure for any purpose you have consented to.

This study may involve unpredictable risks to the participants.

## 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs

may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Wenli Liu, at 713-745-4469) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- This study or your participation in it may be changed or stopped without your consent at any time by the study chair, MD Anderson Cancer Center, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

## **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson, and/or shared with other researchers and/or institutions for use in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD

Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

## Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form
- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## **CONSENT/AUTHORIZATION**

consent form for this study, or have had it read to me. I have had a chance to think about

I understand the information in this consent form. I have had a chance to read the

| it, ask questions, and talk about it with others as needed to enroll me on this study. By signing this consent form, legal rights. I will be given a signed copy of this consent | I am not giving up any of my |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out wher capacity to legally consent to take part in the study and/o own behalf. | • • |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPAN WITNESS TO CONSENT I was present during the explanation of the research to b 2020-0234. | |
| SIGNATURE OF WITNESS TO THE VERBAL CONSEN PRESENTATION (OTHER THAN PHYSICIAN OR STUE A witness signature is only required for vulnerable adult participants of a pediatric participant, leave this line blank and sign on the witness | DY CHAIR)<br>. If witnessing the assent |
| PRINTED NAME OF WITNESS TO THE VERBAL CONS | SENT |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant representative, using language that is understandable ar have fully informed this participant of the nature of this st risks and that the participant understood this explanation | nd appropriate. I believe that I<br>audy and its possible benefits and |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | _ |

| TRA | NSL | .AT | OR |
|-----|-----|-----|----|

| I have translated the above in subtractions) into | nformed consent as written (without additions or<br>and assisted the people | |
|---|---|---|
| , | ame of Language) | 1 1 |
| • | ent by translating all questions and res | ponses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) | | |
| SIGNATURE OF WITNESS (OTHER THAN TRANSLATO OR STUDY CHAIR) | TO THE VERBAL TRANSLATION DR, PARENT/GUARDIAN, | DATE |
| PRINTED NAME OF WITNE | SS TO THE VERBAL TRANSLATION | |